CLINICAL TRIAL: NCT04446364
Title: Ethanolic Extract of Aloe Vera Versus Chlorohexidine as Cavity Disinfectant: A Split-mouth Randomized Clinical Trial
Brief Title: Ethanolic Extract of Aloe Vera Versus Chlorohexidine as Cavity Disinfectant.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Ibrahim Ahmed Hedia, Master degree studnet, Conservative Dentistry Department, Faculty of Dentistry, Cairo University., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ethanolic Extract of Aloe vera
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aloe vera group (Experimental): Gel cavity disinfection
  Interventions: Other: Ethanolic extract of Aloe vera gel cavity disinfectant; Other: Chlorohexadine
- Chlorohexidine group (Active Comparator): 2% cavity disinfection
  Interventions: Other: Ethanolic extract of Aloe vera gel cavity disinfectant; Other: Chlorohexadine

INTERVENTIONS:
Other: Ethanolic extract of Aloe vera gel cavity disinfectant — Application of Aloe vera gel after partial caries removal then taking dentin bacterial sample to be sure for reduction of bacterial count (streptococcus mutans and Lactobacillus) in deep cavity then add final restoration
  Other Names: Aloe vera
Other: Chlorohexadine — 2%Chlorohexadine add on deep cavity as cavity disinfection after partial caries removal. Pre and post excavation bacterial count to measure bacterial reduction then add final restoration

SUMMARY:
This Randomized Clinical Trial will be conducted to compare the efficacy of ethanolic extract of Aloe vera versus chlorhexidine cavity disinfectant in reducing total bacterial count of Streptococcus mutans (SM) and Lactobacilli (LB).

DETAILED DESCRIPTION:
Dental caries remains to be a major oral health problem afflicting people, young and old, especially in developing and underdeveloped countries. Though dentistry has magically developed with newer materials and newer techniques, dental caries remains a disease of great prevalence.

The prevention and control of caries necessitates the elimination of cariogenic bacteria that produce acids responsible for the decrease of pH and starting the process of demineralization.

While the goal of restorative treatments for dental caries is to remove the infected dentin and fill the area with a suitable restorative material, failure to remove the infected teeth surface totally and achieve complete sterilization of the cavity can lead to microleakage, increased pulp sensitivity, pulpal infection and secondary caries that necessitate replacement of restoration.

Therefore, after removal of the carious dentin it is important to eliminate any remaining bacteria that may be present on the cavity walls, in the smear layer, at the enamel-dentin junction, or in the dentinal tubules. But unfortunately, no definitive and reliable criteria are available to ensure the complete removal of carious tooth structure. Many investigations have shown the presence of bacteria in the dentin even after removal of dye-stainable dentin.

Due to indiscriminate use of antimicrobials more and more pathogens are becoming resistant and posing a serious threat in rendering successful treatment of the diseases. With the rise in bacterial resistance to various synthetic antimicrobial agents, there is a considerable interest and a growing trend in the field.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with at least two occlusal deep carious lesions, one on each side, preferred from the same arch.

  * Age range 20-50 years.
  * Systematically health.
  * Adults who were able to give informed consent.
  * Teeth with radiographic evidence of carious lesion that penetrated at least the inner one half of the dentin thickness.

Exclusion Criteria:

* • Patients with clinical and radiographic signs of pulpal involvement.

  * Patients unable to return for recall appointments.
  * Inability of a patient to give informed consent.
  * Teeth with clinical and radiographic sign of pulpal involvement.
  * Teeth where isolation with a rubber dam was not possible

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Bacterial reduction | one year
  Reduction of total bacterial count of SM and LB. IT will be measured before and after cavity disinfectant.

SECONDARY OUTCOMES:
Pulp vitality | one year
  Pulp should be vital instead of death of pulp and loose its vitality

IPD SHARING:
Plan to Share IPD: No